CLINICAL TRIAL: NCT02895386
Title: A Prospective, Randomized, Adaptive, Double-Blind, Sham-Controlled, Multicenter Study to Evaluate the ROX Coupler in Subjects With Hypertension
Brief Title: A Multicenter Study to Evaluate the ROX Coupler in Subjects With Hypertension
Acronym: CONTROL HTN-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company/Sponsor has discontinued business
Sponsor: ROX Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: US HTN-01
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Hypertension; High Blood Pressure
Keywords: Hypertension; High Blood Pressure; Systolic Blood Pressure; Uncontrolled Hypertension; Essential Hypertension; Resistant Hypertension; Vascular Disease
MeSH Terms: conditions — Hypertension; Essential Hypertension; Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment Group A (Active Comparator): ROX Coupler implantation and continuing antihypertensive medications.
  Interventions: Device: ROX Coupler
- Control Group B (Sham Comparator): Sham procedure and continuing current antihypertensive medications.
  Interventions: Other: Sham procedure

INTERVENTIONS:
Device: ROX Coupler — ROX Coupler will be used to create an anastomosis in the iliac region (between the iliac artery and vein).
  Arms: Treatment Group A
Other: Sham procedure — Sham procedure + continuing current antihypertensive medications.
  Arms: Control Group B

SUMMARY:
To evaluate the safety and effectiveness of the ROX Coupler used to create an arteriovenous anastomosis in the iliac region (between the iliac artery and vein) in subjects with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Mean 24-hour ambulatory blood pressure monitoring (ABPM) SBP ≥ 140 mmHg at screening.

Exclusion Criteria:

* Any serious medical condition that may adversely affect the patient's safety, limit the subject's ability to participate in the study, comply with follow-up requirements or impact the scientific integrity of the study.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in mean 24-hour Ambulatory Blood Pressure Monitor systolic blood pressure | Baseline, 6 months
  Change in mean 24-hour Ambulatory Blood Pressure Monitor systolic blood pressure at six month as compared to Baseline

SECONDARY OUTCOMES:
Change in mean office systolic blood pressure | Baseline, 6 months
  Change in mean office systolic blood pressure at six months as compared to Baseline

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Cardiology P.C. Research, Birmingham, Alabama
  - UAB Division of Cardiovascular Disease, Birmingham, Alabama
  - The Cardiac and Vascular Institute Research Foundation, Gainesville, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Cardiology Associates Research, Tupelo, Mississippi
  - Northwell Health - North Shore University Hospital, Manhasset, New York
  - Northwell Health - Lenox Hill Hospital, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - CAMC Clinical Trials Center, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lobo MD, Sobotka PA, Stanton A, Cockcroft JR, Sulke N, Dolan E, van der Giet M, Hoyer J, Furniss SS, Foran JP, Witkowski A, Januszewicz A, Schoors D, Tsioufis K, Rensing BJ, Scott B, Ng GA, Ott C, Schmieder RE; ROX CONTROL HTN Investigators. Central arteriovenous anastomosis for the treatment of patients with uncontrolled hypertension (the ROX CONTROL HTN study): a randomised controlled trial. Lancet. 2015 Apr 25;385(9978):1634-41. doi: 10.1016/S0140-6736(14)62053-5. Epub 2015 Jan 23. PMID 25620016
- [Background] Lobo MD, Ott C, Sobotka PA, Saxena M, Stanton A, Cockcroft JR, Sulke N, Dolan E, van der Giet M, Hoyer J, Furniss SS, Foran JP, Witkowski A, Januszewicz A, Schoors D, Tsioufis K, Rensing BJ, Scott B, Ng GA, Schmieder RE. Central Iliac Arteriovenous Anastomosis for Uncontrolled Hypertension: One-Year Results From the ROX CONTROL HTN Trial. Hypertension. 2017 Dec;70(6):1099-1105. doi: 10.1161/HYPERTENSIONAHA.117.10142. Epub 2017 Oct 23. PMID 29061728
- See also: Corporate website — http://www.roxmedical.com